CLINICAL TRIAL: NCT02811835
Title: Renal Sensing of the Acidifying Effect of Sulphur-containing Amino Acids: Consequences for the Relation Between Protein Intake and Blood Pressure in Renal Transplant Recipients
Brief Title: TransplantLines Food and Nutrition Biobank and Cohort Study (TxL-FN)
Acronym: TxL-FN
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Stephan J.L. Bakker, Prof. dr., University Medical Center Groningen
Other Study IDs: METc2008/186
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Transplantation Infection; Renal Transplant Donor of Left Kidney

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples Without DNA — Serum and EDTA plasma stored at -80 degrees Centigrade Vials from 24h urine samples stored at -80 degrees Centigrade
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Renal Transplant Recipients: Renal Transplant Recipients that were more than 1 year post-transplantation
- Healthy Controls: Healthy subjects being evaluated as potential living kidney donors

SUMMARY:
Short-term (1-year) results of renal transplantation are now excellent (over 95%). Long-term (10-year and longer) results are, however, still disappointing. Where most research has focused on immunosuppression and infections, the investigators hypothesize that due to poor homeostatic capacity and necessary use of immunosuppressive and other drugs, renal transplant recipients are much more susceptible to poor dietary habits and exposure to potentially toxic contaminants than people of the general population, and that this contributes to accelerated function loss of the graft and excess risk of premature mortality, both contributing to poor long-term results. This study is a biobank and cohort study which investigates this hypothesis.

DETAILED DESCRIPTION:
Short-term (1-year) results of renal transplantation are now excellent (over 95%). Long-term (10-year and longer) results are, however, still disappointing. Where most research has focused on immunosuppression and infections, the investigators hypothesize that due to poor homeostatic capacity and necessary use of immunosuppressive and other drugs, renal transplant recipients are much more susceptible to poor dietary habits and exposure to potentially toxic contaminants than people of the general population, and that this contributes to accelerated function loss of the graft and excess risk of premature mortality, both contributing to poor long-term results.

To investigate one part of this overarching hypothesis, the investigators wrote a project on around the specific topic of the relation between dietary acid load, ammoniagenesis and its potential influence on blood pressure. The investigators used this project to build a biobank and cohort in which they can test additional hypotheses on the relation between diet, contaminants and development of graft failure and the occurrence of mortality.

The investigators also included 300 healthy controls to compare diet, contaminant exposure and biomarkers with the renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria: More than one year after transplantation, prognosis > 1 year, stable outpatients situation -

Exclusion Criteria: Acute illnesses, fever, current hospitalisation

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Renal Transplant Recipients and Healthy Potential Kidney Donors
Sampling Method: Non-Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Graft failure | 20 years
  Return to dialysis or re-transplantation
All-cause mortality | 20 years
  Death

SECONDARY OUTCOMES:
Cardiovascular mortality | 20 years
  Cause specific mortality
Cancer mortality | 20 years
  Cause specific mortality
Infectious disease mortality | 20 years
  Cause specific mortality

OTHER OUTCOMES:
Change in renal function | 20 years
  Change in renal function over time
New Onset Diabetes After Transplantation | 20 years
  New Onset Diabetes

IPD SHARING:
Plan to Share IPD: Yes
Each participant has a study number which is not traceable to the patient in the study

REFERENCES:
- [Derived] Kremer D, Rawee P, Knobbe TJ, Vinke JSJ, Luersen K, Leaf DE, Swinkels DW, de Borst MH, Rimbach G, Bakker SJL, Eisenga MF. Higher Urinary Iron Levels Are Associated with Kidney Dysfunction, Tubular Damage, and Increased Mortality in Kidney Transplant Recipients. Kidney360. 2025 Nov 1;6(11):1970-1980. doi: 10.34067/KID.0000000878. Epub 2025 Jun 26. PMID 40569672
- [Derived] Post A, Groothof D, Kremer D, Knobbe TJ, Abma W, Koops CA, Tsikas D, Wallimann T, Dullaart RPF, Franssen CFM, Kema IP, Heiner-Fokkema MR, Bakker SJL. Creatine homeostasis and the kidney: comparison between kidney transplant recipients and healthy controls. Amino Acids. 2024 Jun 13;56(1):42. doi: 10.1007/s00726-024-03401-w. PMID 38869518
- [Derived] Post A, Kremer D, Groothof D, Seidel U, Huebbe P, Franssen CFM, Kema IP, Luersen K, Rimbach G, Bakker SJL. Dietary lithium intake, graft failure and mortality in kidney transplant recipients. Nephrol Dial Transplant. 2023 Jul 31;38(8):1867-1879. doi: 10.1093/ndt/gfac340. PMID 36564033
- [Derived] Kremer D, Alkaff FF, Post A, Knobbe TJ, Tepel M, Thaunat O, Berger SP, van den Born J, Genovese F, Karsdal MA, Rasmussen DGK, Bakker SJL. Plasma endotrophin, reflecting tissue fibrosis, is associated with graft failure and mortality in KTRs: results from two prospective cohort studies. Nephrol Dial Transplant. 2023 Mar 31;38(4):1041-1052. doi: 10.1093/ndt/gfac332. PMID 36535643
- [Derived] Oste MCJ, Duan MJ, Gomes-Neto AW, Vinke PC, Carrero JJ, Avesani C, Cai Q, Dekker LH, Navis GJ, Bakker SJL, Corpeleijn E. Ultra-processed foods and risk of all-cause mortality in renal transplant recipients. Am J Clin Nutr. 2022 Jun 7;115(6):1646-1657. doi: 10.1093/ajcn/nqac053. PMID 35470855
- [Derived] Kremer D, Post A, Gomes-Neto AW, Groothof D, Kunutsor SK, Nilsen T, Hidden C, Sundrehagen E, Eisenga MF, Navis G, Bakker SJL; TransplantLines Investigators. Plasma neutrophil gelatinase-associated lipocalin and kidney graft outcome. Clin Kidney J. 2021 Nov 8;15(2):235-243. doi: 10.1093/ckj/sfab219. eCollection 2022 Feb. PMID 35145638
- [Derived] Stam SP, Sokooti S, Eisenga MF, van der Veen A, Gomes-Neto AW, van Dijk PR, van Zanden JJ, Vos MJ, Kema IP, van Beek AP, Bakker SJL; TransplantLines Investigators. Androgens and Development of Posttransplantation Diabetes Mellitus in Male Kidney Transplant Recipients: A Post Hoc Analysis of a Prospective Study. Diabetes Care. 2021 Dec;44(12):2683-2690. doi: 10.2337/dc21-0237. Epub 2021 Oct 5. PMID 34610923
- [Derived] Yeung SMH, Gomes-Neto AW, Oste MCJ, van den Berg E, Kootstra-Ros JE, Sanders JSF, Berger SP, Carrero JJ, De Borst MH, Navis GJ, Bakker SJL. Net Endogenous Acid Excretion and Kidney Allograft Outcomes. Clin J Am Soc Nephrol. 2021 Sep;16(9):1398-1406. doi: 10.2215/CJN.00780121. Epub 2021 Jun 16. PMID 34135022
- [Derived] Cai Q, Oste MCJ, Gomes-Neto AW, Dekker LH, Borgonjen-van den Berg KJ, Geleijnse JM, Bakker SJL, de Borst MH, Navis GJ. Metabolic syndrome-related dietary pattern and risk of mortality in kidney transplant recipients. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1129-1136. doi: 10.1016/j.numecd.2021.01.005. Epub 2021 Jan 19. PMID 33618925
- [Derived] Klont F, Kremer D, Gomes Neto AW, Berger SP, Touw DJ, Hak E, Bonner R, Bakker SJL, Hopfgartner G. Metabolomics data complemented drug use information in epidemiological databases: pilot study of potential kidney donors. J Clin Epidemiol. 2021 Jul;135:10-16. doi: 10.1016/j.jclinepi.2021.02.008. Epub 2021 Feb 9. PMID 33577985
- [Derived] Sotomayor CG, Oskooei SS, Bustos NI, Nolte IM, Gomes-Neto AW, Erazo M, Gormaz JG, Berger SP, Navis GJ, Rodrigo R, Dullaart RPF, Bakker SJL. Serum uric acid is associated with increased risk of posttransplantation diabetes in kidney transplant recipients: a prospective cohort study. Metabolism. 2021 Mar;116:154465. doi: 10.1016/j.metabol.2020.154465. Epub 2020 Dec 13. PMID 33316268
- [Derived] Post A, Said MY, Gomes-Neto AW, Minovic I, Groothof D, Swarte JC, Boer T, Kema IP, Heiner-Fokkema MR, Franssen CFM, Bakker SJL. Urinary 3-hydroxyisovaleryl carnitine excretion, protein energy malnutrition and risk of all-cause mortality in kidney transplant recipients: Results from the TransplantLines cohort studies. Clin Nutr. 2021 Apr;40(4):2109-2120. doi: 10.1016/j.clnu.2020.09.035. Epub 2020 Oct 1. PMID 33071013
- [Derived] Sotomayor CG, Groothof D, Vodegel JJ, Eisenga MF, Knobbe TJ, IJmker J, Lammerts RGM, de Borst MH, Berger SP, Nolte IM, Rodrigo R, Slart RHJA, Navis GJ, Touw DJ, Bakker SJL. Plasma cadmium is associated with increased risk of long-term kidney graft failure. Kidney Int. 2021 May;99(5):1213-1224. doi: 10.1016/j.kint.2020.08.027. Epub 2020 Sep 14. PMID 32941876
- [Derived] Douwes RM, Gomes-Neto AW, Eisenga MF, Van Loon E, Schutten JC, Gans ROB, Naesens M, van den Berg E, Sprangers B, Berger SP, Navis G, Blokzijl H, Meijers B, Bakker SJL, Kuypers D. The association between use of proton-pump inhibitors and excess mortality after kidney transplantation: A cohort study. PLoS Med. 2020 Jun 15;17(6):e1003140. doi: 10.1371/journal.pmed.1003140. eCollection 2020 Jun. PMID 32542023
- [Derived] Vulto A, Minovic I, de Vries LV, Timmermans AC, van Faassen M, Gomes Neto AW, Touw DJ, de Jong MFC, van Beek AP, Dullaart RPF, Navis G, Kema IP, Bakker SJL. Endogenous urinary glucocorticoid metabolites and mortality in prednisolone-treated renal transplant recipients. Clin Transplant. 2020 Apr;34(4):e13824. doi: 10.1111/ctr.13824. Epub 2020 Mar 3. PMID 32052523
- [Derived] Gomes-Neto AW, Oste MCJ, Sotomayor CG, van den Berg E, Geleijnse JM, Berger SP, Gans ROB, Bakker SJL, Navis GJ. Mediterranean Style Diet and Kidney Function Loss in Kidney Transplant Recipients. Clin J Am Soc Nephrol. 2020 Feb 7;15(2):238-246. doi: 10.2215/CJN.06710619. Epub 2020 Jan 2. PMID 31896540
- [Derived] Gomes-Neto AW, Oste MCJ, Sotomayor CG, V D Berg E, Geleijnse JM, Gans ROB, Bakker SJL, Navis GJ. Fruit and Vegetable Intake and Risk of Posttransplantation Diabetes in Renal Transplant Recipients. Diabetes Care. 2019 Sep;42(9):1645-1652. doi: 10.2337/dc19-0224. Epub 2019 Jul 11. PMID 31296643
- [Derived] Oste MCJ, Gomes-Neto AW, Corpeleijn E, Gans ROB, de Borst MH, van den Berg E, Soedamah-Muthu SS, Kromhout D, Navis GJ, Bakker SJL. Dietary Approach to Stop Hypertension (DASH) diet and risk of renal function decline and all-cause mortality in renal transplant recipients. Am J Transplant. 2018 Oct;18(10):2523-2533. doi: 10.1111/ajt.14707. Epub 2018 Mar 23. PMID 29464830
- [Derived] Minovic I, van der Veen A, van Faassen M, Riphagen IJ, van den Berg E, van der Ley C, Gomes-Neto AW, Geleijnse JM, Eggersdorfer M, Navis GJ, Kema IP, Bakker SJ. Functional vitamin B-6 status and long-term mortality in renal transplant recipients. Am J Clin Nutr. 2017 Dec;106(6):1366-1374. doi: 10.3945/ajcn.117.164012. Epub 2017 Oct 4. PMID 28978540
- [Derived] Minovic I, Riphagen IJ, van den Berg E, Kootstra-Ros JE, van Faassen M, Gomes Neto AW, Geleijnse JM, Gans RO, Eggersdorfer M, Navis GJ, Kema IP, Bakker SJ. Vitamin B-6 deficiency is common and associated with poor long-term outcome in renal transplant recipients. Am J Clin Nutr. 2017 Jun;105(6):1344-1350. doi: 10.3945/ajcn.116.151431. Epub 2017 May 3. PMID 28468895
- [Derived] Eisenga MF, Kieneker LM, Soedamah-Muthu SS, van den Berg E, Deetman PE, Navis GJ, Gans RO, Gaillard CA, Bakker SJ, Joosten MM. Urinary potassium excretion, renal ammoniagenesis, and risk of graft failure and mortality in renal transplant recipients. Am J Clin Nutr. 2016 Dec;104(6):1703-1711. doi: 10.3945/ajcn.116.134056. Epub 2016 Nov 9. PMID 27935524